CLINICAL TRIAL: NCT07356700
Title: Deciphering the Factors of Longevity Through a Multi-Omics Study in Long-Lived Individuals in Hong Kong
Status: Not yet recruiting | Type: Observational
Sponsor: Hong Kong University of Science and Technology (Other)
Collaborators: Hong Kong Center for Neurodegenerative Diseases (Other)
Responsible Party: Principal Investigator, Hiu Yi Wong, Research Assistant Professor, Hong Kong University of Science and Technology
Other Study IDs: HREP-2025-0294
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aging
Keywords: Aging; Multi-omics; AI-based tool; Longevity
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- long-lived individuals (LLIs): individuals aged 95 years or older
  Interventions: Other: Observational
- Elderly controls: elderly people aged 65-94 years
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Clinical profile, blood collection, cognitive assessment, questionnaires on modifiable risk factors

SUMMARY:
Population aging is changing societal dynamics and poses significant global challenges. By 2050, an estimated 1.6 billion people worldwide will be over age 65. Because aging is the primary risk factor for many common chronic diseases, it is essential to reduce the burden of age-related illnesses and promote healthy aging. Hong Kong has one of the largest proportions of elderly adults and has the highest life expectancy in the world, with approximately 11,575 centenarians reported in 2021. Thus, the long-lived population in Hong Kong is a valuable resource for studying healthy aging.

Longevity is a complex trait influenced by genetic, environmental, and behavioral factors. To unveil the mechanisms leading to longevity and healthy aging, researchers focused on centenarians who are extremely long living. Comparisons between long-lived individuals (LLIs) and others have identified several genetic factors and protein markers associated with longevity. Previous centenarian studies revealed that centenarians and their offsprings have a 5-fold lower risk of developing age-related diseases such as Alzheimer's disease and higher cognitive reserve. Certain protein signatures predict longer survival and centenarians acquire aging signatures much later than elderly in the general population. Certain healthy lifestyle leads to higher chance becoming centenarians, including never smoking, exercise and greater dietary diversity.

Despite emerging studies on centenarian population, an integrated approach to understand diverse molecular signatures of longevity is still lacking. Moreover, most of the centenarian studies are based on European descents. To conclude, a multi-omics study examining the genetic, proteomic, metabolomic, and microbiota profiles of LLIs in Chinese population is necessary.

Hence, the study proposed herein aims to identify multi-omics biomarkers that can be used to monitor aging processes and related diseases. In addition, it will provide candidate modifiable factors to promote healthy aging, focusing on Chinese population and local Hong Kong population for the first time. Ultimately, the insights gained from this research will inform the development of effective strategies to enhance healthy aging and improve the quality of life of our local aging population.

DETAILED DESCRIPTION:
The proposed research is a cross-sectional study that will last for 5 years. 500 individuals aged 95 years or older (i.e., LLIs) from various communities in Hong Kong will be recruited. LLIs will be recruited through advertisements as well as collaboration with geriatric community centers and non-government organizations (NGOs). Participants will be recruited at geriatric centers and NGOs to collect demographic information, family history, medical history, and medication records. Blood samples for clinical chemistry and multi-omics study will be collected. Furthermore, cognitive and functional assessment using various scoring systems will be performed to assess cognition and activities of daily living.

In addition, a control cohort of elderly people (aged 65-94 years, n = 2,000) based on our in-house Alzheimer's disease registry and community cohort will be developed. Accordingly, demographics, clinical profiles, cognitive and functional scores, and multi-omics data between the LLI and control cohorts will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Han Chinese ethnicity
2. Able to provide official evidence for being 95 years or older (e.g., a birth certificate)
3. Mentally capable of consenting to join the study with or without informant presence
4. Consent to donation of biospecimens (i.e., blood)

Exclusion Criteria:

1. Mentally incapable of consenting to join the study even with the presence of an informant
2. Refusal to provide blood samples

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly with extreme longevity (aged >=95 years old)
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Biobank of LLIs | 3-5 years
  A comprehensive cohort of LLIs with data on demographics, clinical profiles, cognitive and functional assessments, lifestyle, and genomic and proteomic biomarkers
Genetic and modifiable factors associated with longevity | 3-5 years
  Genetic and modifiable factors associated with longevity

SECONDARY OUTCOMES:
AI-based model | 5 years
  AI-based model to elucidate candidate modifiable factors that promote healthy aging
Healthy aging strategies | 5 years
  Recommendations for personalized strategies to enhance healthy aging in the elderly population

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ip, PhD, Principal Investigator — Hong Kong University of Science and Technology
Locations (1):
- Hong Kong University of Science and Technology, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Wang K, Jigeer G, Jensen G, Tucker KL, Lv Y, Shi X, Gao X. Healthy Lifestyle and the Likelihood of Becoming a Centenarian. JAMA Netw Open. 2024 Jun 3;7(6):e2417931. doi: 10.1001/jamanetworkopen.2024.17931. PMID 38900423
- [Background] Sebastiani P, Federico A, Morris M, Gurinovich A, Tanaka T, Chandler KB, Andersen SL, Denis G, Costello CE, Ferrucci L, Jennings L, Glass DJ, Monti S, Perls TT. Protein signatures of centenarians and their offspring suggest centenarians age slower than other humans. Aging Cell. 2021 Feb;20(2):e13290. doi: 10.1111/acel.13290. Epub 2021 Jan 29. PMID 33512769
- [Background] Holstege H, Beker N, Dijkstra T, Pieterse K, Wemmenhove E, Schouten K, Thiessens L, Horsten D, Rechtuijt S, Sikkes S, van Poppel FWA, Meijers-Heijboer H, Hulsman M, Scheltens P. The 100-plus Study of cognitively healthy centenarians: rationale, design and cohort description. Eur J Epidemiol. 2018 Dec;33(12):1229-1249. doi: 10.1007/s10654-018-0451-3. Epub 2018 Oct 25. PMID 30362018
- [Background] Zhang M, Ganz AB, Rohde S, Rozemuller AJM, Bank NB, Reinders MJT, Scheltens P, Hulsman M, Hoozemans JJM, Holstege H. Resilience and resistance to the accumulation of amyloid plaques and neurofibrillary tangles in centenarians: An age-continuous perspective. Alzheimers Dement. 2023 Jul;19(7):2831-2841. doi: 10.1002/alz.12899. Epub 2022 Dec 30. PMID 36583547
- [Background] Tesi N, van der Lee S, Hulsman M, van Schoor NM, Huisman M, Pijnenburg Y, van der Flier WM, Reinders M, Holstege H. Cognitively healthy centenarians are genetically protected against Alzheimer's disease. Alzheimers Dement. 2024 Jun;20(6):3864-3875. doi: 10.1002/alz.13810. Epub 2024 Apr 18. PMID 38634500
- [Background] Hong Kong Centenarian Study 2 Project Report, 2023, Hong Kong Shue Yan University
- [Background] 2021 Thematic Report: Older Persons, HKSAR Census and Statistics Department